CLINICAL TRIAL: NCT03116152
Title: Efficacy and Safety Evaluation of IBI308 Versus Paclitaxel/Irinotecan in Patients With Advanced/Metastatic Esophageal Squamous Cell Carcinoma After Failure of First-line Treatment: a Randomized, Open-label, Multicenter, Phase 2 Study (ORIENT-2)
Brief Title: Study of IBI308 With Advanced/Metastatic Esophageal Squamous Cell Carcinoma After Failure of First-line Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308A201
Record Dates: First submitted 2017-03-15; First posted 2017-04-14 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab; Paclitaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI308 (Experimental): IBI308 200mg Intravenous drip every three weeks
  Interventions: Biological: IBI308
- paclitaxel/irinotecan (Active Comparator): paclitaxel 175mg/㎡ Intravenous drip every three weeks； irinotecan 180mg/㎡ Intravenous drip every two weeks
  Interventions: Drug: paclitaxel/ irinotecan

INTERVENTIONS:
Biological: IBI308 — IBI308 200mg Intravenous drip every three weeks；
  Arms: IBI308
Drug: paclitaxel/ irinotecan — paclitaxel 175mg/㎡ Intravenous drip every three weeks or irinotecan 180mg/㎡ Intravenous drip every two weeks
  Arms: paclitaxel/irinotecan

SUMMARY:
Efficacy and safety evaluation of IBI308 versus paclitaxel/irinotecan in patients with advanced/metastatic esophageal squamous cell carcinoma after failure of first-line treatment: a randomized, open-label, multicenter, phase 2 study

DETAILED DESCRIPTION:
Efficacy and safety evaluation of IBI308 versus paclitaxel/irinotecan in patients with advanced/metastatic esophageal squamous cell carcinoma after failure of first-line treatment: a randomized, open-label, multicenter, phase 2 study (ORIENT-2)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced unresectable or metastatic esophageal squamous cell carcinoma (excluding mixed adenosquamous carcinoma and other pathological types).
2. Imaging evidence (e.g. CT scan) or clinical evidence (e.g. cytological report of new ascites or pleural effusion) of disease progression during or after first-line chemotherapy; Subjects have to receive at least one dose of first-line treatment, permitting discontinuation or dose reduction of one drug or exchange of fluorouracil drugs used during first-line treatment, and patients discontinuing first-line treatment due to intolerable toxicity are allowed to be enrolled; Neoadjuvant or adjuvant therapy (chemotherapy or chemo-radiotherapy) should be regarded as first-line treatment if there is disease progression during treatment or within 6 months after treatment discontinuation.
3. At least one measurable lesion according to RECIST v1.1.
4. ECOG PS score of 0 or 1.
5. Subjects who have signed the written informed consent form and are able to follow the visit schedule and relevant procedures as specified in the study protocol.
6. Age ≥ 18 and ≤ 75 years.
7. Life expectancy ≥ 12 weeks.
8. Female subjects of childbearing potential or male subjects with sexual partners of childbearing potential should use effective contraception throughout and within 6 months after treatment.
9. Adequate organ and bone marrow functions, defined as follows:

   * Hematology: absolute neutrophil count (ANC) ≥ 1.5×10^9/L; Platelet (PLT) count ≥ 100×10^9/L; Hemoglobin (HGB) ≥ 9.0 g/dL.
   * Liver function: serum total bilirubin (TBIL) ≤ 1.5×upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; Serum albumin ≥ 28 g/L.
   * Renal function: Serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance (Ccr) ≥ 40 mL/min (calculated using the standard Cockcroft -Gault formula):

     * Females: CrCl = (140-age) x body weight (kg) x 0.85/(72 x serum creatinine (mg/dL))
     * Males: CrCl = (140-age) x body weight (kg) x 1.00/(72 x serum creatinine (mg/dL))

Exclusion Criteria:

1. Prior exposure to any anti-PD-1 or anti-PD-L1 antibody.
2. Concurrent participation in another interventional clinical study, except for observational (non-interventional) clinical studies or in the follow-up phase of an interventional study.
3. Receipt of any investigational products within 4 weeks prior to the first dose of study treatment.
4. Receipt of the last dose of anti-tumor therapy (chemotherapy, targeted therapy, tumor immunotherapy, tumor embolization) within 3 weeks prior to the first dose of study treatment.
5. Radiotherapy within 4 weeks prior to the first dose of study treatment.
6. Receipt of immunosuppressive agents within 4 weeks prior to the first dose of study treatment, excluding topical glucocorticoids for intranasal, inhalation or other routes of administration, or physiological doses of systemic glucocorticoids (i.e., no more than 10 mg/day prednisone or equivalent doses of other glucocorticoids).
7. Receipt of a live attenuated vaccine within 4 weeks prior to the first dose of study treatment or planned receipt of a live attenuated vaccine during the study.
8. Subjects who have undergone major surgical procedures (craniotomy, thoracotomy or laparotomy) within 4 weeks prior to the first dose of study treatment or have unhealed wound, ulcers or bone fracture.
9. Presence of toxicities induced by previous anti-tumor therapy that have not recovered to Grade 0 or 1 as assessed per NCI CTCAE 4.03 (National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03) prior to the first dose of study treatment, excluding alopecia, and non-clinically significant and asymptomatic laboratory abnormalities.
10. Known symptomatic metastases to central nervous system (CNS) and/or carcinomatous meningitis. Subjects previously treated for brain metastasis are eligible for the study provided the brain metastasis has remained stable for at least 4 weeks before first dose of study treatment; Neurological symptoms must be recovered to grade 0 or 1 as per NCI CTCAE version 4.03.
11. Active, known or suspected autoimmune diseases (refer to Appendix 6) or a history of such disease in the past 2 years (patients with vitiligo, psoriasis, alopecia or Grave's disease requiring no systemic treatment in the past 2 years, patients with hypothyroidism requiring only thyroid hormone replacement therapy and patients with type I diabetes requiring only insulin replacement therapy can be enrolled).
12. Known history of primary immunodeficiency.
13. Known active tuberculosis (TB).
14. Known history of allotransplantation and allogeneic hematopoietic stem cell transplantation.
15. Known hypersensitivity to any component of the monoclonal antibody, paclitaxel or irinotecan formulation.
16. Uncontrolled concurrent diseases, including but not limited to:

    * HIV infection (HIV antibody positive).
    * Active or clinically uncontrolled severe infections.
    * Symptomatic congestive heart failure (New York Heart Association Class II-IV) or symptomatic or poorly controlled arrhythmia.
    * Uncontrolled arterial hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg) despite standard treatment.
    * Any arterial thromboembolism events within 6 months prior to inclusion for treatment, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attacks.
    * Significant malnutrition, if intravenous nutrient solution supplement is required; Except for malnutrition corrected for more than 4 weeks before first dose of study treatment.
    * Tumor invasion into surrounding vital organs (e.g., aorta and trachea) or a risk for esophagotracheal fistula or esophagopleural fistula.
    * Post esophageal or intratracheal stenting.
    * History of deep vein thrombosis (DVT), pulmonary embolism, or any other serious thromboembolism within 3 months prior to enrollment (implanted venous access port or catheter-related thrombosis, or superficial venous thrombosis is not considered as "serious"thromboembolism).
    * Uncontrolled metabolic disorders or other non-malignant organic or systemic diseases or reactions secondary to cancer, which can result in high medical risks and/or uncertainty in survival evaluations.
    * Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh class B or even more severe cirrhosis.
    * History of intestinal obstruction or the following diseases: inflammatory bowel disease or extensive bowel resection (partial colectomy or extensive resection of the small intestine, concurrent chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
    * Other acute or chronic diseases, mental disorders or abnormal laboratory findings that may lead to the following results: increase risks associated with study participation in the study or use of the study drug, or interfere with the interpretation of study results, and render the patient ineligible for the study at the investigator's discretion.
17. Known acute or chronic active hepatitis B (HBsAg positive and HBV DNA ≥200 IU/mL or ≥ 10^3 copies/mL) or acute or chronic active hepatitis C (HCV antibody positive and positive for HCV RNA test).
18. History of gastrointestinal perforation and/or fistula within 6 months prior to study inclusion.
19. Presence of interstitial lung disease.
20. Clinically uncontrollable effusion of the third space, such as pleural effusion and ascites that can not be controlled by drainage or other methods before enrollment.
21. History of other primary malignancies, excluding:

    * A malignancy with complete remission for at least 2 years before enrollment and requiring no other treatment during the study;
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of relapse;
    * Adequately treated carcinoma in situ without evidence of relapse.
22. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of PLA Ceneral Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu J, Li Y, Fan Q, Shu Y, Yang L, Cui T, Gu K, Tao M, Wang X, Cui C, Xu N, Xiao J, Gao Q, Liu Y, Zhang T, Bai Y, Li W, Zhang Y, Dai G, Ma D, Zhang J, Bai C, Huang Y, Liao W, Wu L, Chen X, Yang Y, Wang J, Ji S, Zhou H, Wang Y, Ma Z, Wang Y, Peng B, Sun J, Mancao C. Clinical and biomarker analyses of sintilimab versus chemotherapy as second-line therapy for advanced or metastatic esophageal squamous cell carcinoma: a randomized, open-label phase 2 study (ORIENT-2). Nat Commun. 2022 Feb 14;13(1):857. doi: 10.1038/s41467-022-28408-3. PMID 35165274

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 253 enrolled. 190 randomized. Non-randomized reasons: 55 no longer met study criteria, 4 withdrew consent, 4 other. 181 treated (94 sintilimab, 87 chemotherapy).
Groups:
- Sintilimab: Sintilimab (IBI308) 200mg Intravenous drip every three weeks
- Chemotherapy: paclitaxel 175mg/㎡ Intravenous drip every three weeks； irinotecan 180mg/㎡ Intravenous drip every two weeks
Period: Overall Study
Arm/Group | Sintilimab | Chemotherapy
Started | 95 | 95
Treated (The number of participants who were treated after randomization) | 94 | 87
Completed | 4 | 0
Not Completed | 91 | 95
Not completed — Disease Progression | 49 | 47
Not completed — Death | 5 | 2
Not completed — Adverse Event | 21 | 7
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 3 | 2
Not completed — other | 11 | 34

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Sintilimab | Chemotherapy | Total
Number analyzed (Participants) | 95 | 95 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 75 | 149
  >=65 years | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (7.23) | 59.4 (7.06) | 59.1 (7.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 88 | 84 | 172
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 95 | 95 | 190
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 95 | 95 | 190

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: OS was defined as the time from randomization to death due to any cause. Median OS in all participants is presented.
Time Frame: Through Final Analysis data cutoff date of 2-August-2019 (up to approximately 26 months)
Population: The efficacy analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Sintilimab | Chemotherapy
Number analyzed (Participants) | 95 | 95
month | 7.23 [5.82 to 9.69] | 6.21 [5.39 to 7.85]
Statistical Analysis 1: Comparison: Sintilimab vs Chemotherapy; Test type: Superiority; p = 0.032, Log Rank; Hazard Ratio (HR) = 0.701, 95% CI 2-sided [0.504 to 0.972]

2. Secondary Outcome: Progression-free Survival
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) as determined by the investigator, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Unequivocal progression of non-target leisions and the appearance of ≥1 new lesions were also considered as PD.
Time Frame: Through Final Analysis data cutoff date of 2-August-2019 (up to approximately 26 months)
Population: The efficacy analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Sintilimab | Chemotherapy
Number analyzed (Participants) | 95 | 95
month | 1.58 [1.45 to 2.76] | 2.86 [2.56 to 3.55]
Statistical Analysis 1: Comparison: Sintilimab vs Chemotherapy; Test type: Superiority; p = 0.979, Log Rank; Hazard Ratio (HR) = 1.002, 95% CI 2-sided [0.722 to 1.391]

3. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate (ORR) was defined as the proportion of randomized participants who achieved a best response of complete response (CR) or partial response (PR) using the RECIST1.1 criteria as per investigator assessment.
Time Frame: Through Final Analysis data cut-off date of 2-August-2019 (up to approximately 26 months)
Population: The efficacy analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sintilimab | Chemotherapy
Number analyzed (Participants) | 95 | 95
Percentage of Participants | 12.6 [6.7 to 21.0] | 6.3 [2.4 to 13.2]
Statistical Analysis 1: Comparison: Sintilimab vs Chemotherapy; Test type: Superiority; Difference in Percentages = 6.3, 95% CI 2-sided [-2.2 to 15.4]

4. Secondary Outcome: Duration of Response
Description: Duration of response (DoR) was defined as the time from the date of the first investigator-assessed response (CR or PR) to the date of subsequent investigator-assessed PD or death, whichever is earlier.
Time Frame: Through Final Analysis data cutoff date of 2-August-2019 (up to approximately 26 months)
Population: The efficacy analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Sintilimab | Chemotherapy
Number analyzed (Participants) | 95 | 95
month | 8.28 [2.92 to 20.9] | 6.21 [4.57 to 8.38]
Statistical Analysis 1: Comparison: Sintilimab vs Chemotherapy; Test type: Superiority; p = 0.345, Log Rank

ADVERSE EVENTS:
Time Frame: Through the Analysis data cutoff date of 2-October-2019 (up to approximately 26 months). The cutoff date for the primary efficacy analysis was 02 August 2019 when 150 OS events were actually observed. Upon the observation, the study follow-up was extended for another 2 months. The safety data was cut off as of 2-October-2019. AEs were collected till 90 days after the last dose.
Description: All-Cause Mortality assessed for all the participants who Started the study and Serious and Other (Not Including Serious) Adverse Events were assessed in all participants who received ≥1 dose of study treatment. 181 treated (94 sintilimab, 87chemotherapy).
Arm/Group | Sintilimab | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 73/95 | 82/95
Serious Adverse Events (participants affected / at risk) | 41/94 | 23/87
Other Adverse Events (participants affected / at risk) | 88/94 | 78/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab (N=94) | Chemotherapy (N=87)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastric fistula (Gastrointestinal disorders) | 1 | 0
Gastropleural fistula (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 0
Lung infection (Infections and infestations) | 5 | 4
Biliary tract infection (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiratio (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asphyxia (Reproductive system and breast disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Accidental death (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 6
Cardiac failure (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Amylase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab (N=94) | Chemotherapy (N=87)
Weight decreased (Investigations) | 28 | 15
White blood cell count decreased (Investigations) | 13 | 45
Aspartate aminotransferase increased (Investigations) | 12 | 6
Alanine aminotransferase increased (Investigations) | 10 | 6
Amylase increased (Investigations) | 10 | 1
Lymphocyte count decreased (Investigations) | 11 | 11
Neutrophil count decreased (Investigations) | 10 | 32
Gamma-glutamyltransferase increased (Investigations) | 9 | 3
Platelet count decreased (Investigations) | 9 | 12
Hypoproteinaemia (Metabolism and nutrition disorders) | 23 | 8
Decreased appetite (Metabolism and nutrition disorders) | 14 | 17
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 10 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 10
Hypochloraemia (Metabolism and nutrition disorders) | 9 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 4
Anaemia (Blood and lymphatic system disorders) | 46 | 43
Constipation (Gastrointestinal disorders) | 19 | 14
Nausea (Gastrointestinal disorders) | 12 | 31
Vomiting (Gastrointestinal disorders) | 12 | 21
Diarrhoea (Gastrointestinal disorders) | 12 | 32
Abdominal pain (Gastrointestinal disorders) | 6 | 8
Asthenia (General disorders) | 16 | 23
Pyrexia (General disorders) | 13 | 6
Pain (General disorders) | 5 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Hypothyroidism (Endocrine disorders) | 13 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 10 | 5
Proteinuria (Renal and urinary disorders) | 8 | 8
Lung infection (Infections and infestations) | 7 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 13
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 6
Blood alkaline phosphatase increased (Investigations) | 7 | 2
Blood bilirubin increased (Investigations) | 6 | 3
Lipase increased (Investigations) | 5 | 0
Neutrophil count increased (Investigations) | 6 | 2
White blood cell count increased (Investigations) | 6 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Headache (Nervous system disorders) | 5 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 6
Insomnia (Psychiatric disorders) | 5 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Hypertension (Vascular disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT03116152/Prot_SAP_000.pdf